CLINICAL TRIAL: NCT06260891
Title: Zinc Supplementation in Sickle Cell Disease: A Precursor to the Think Zinc for Bones Trial
Acronym: ZnSCD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Children's Hospital of Philadelphia (Other); University of Pennsylvania (Other); Children's Hospital Medical Center, Cincinnati (Other); American Society of Hematology (Other); Baylor College of Medicine (Other); Thomas Jefferson University (Other); Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: ZnSCD
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Zinc

STUDY DESIGN:
Intervention Model Description: This is a delayed start parallel design where all subjects will have a usual care period, 2 baseline samples 4 weeks apart, followed by a 12 week zinc intervention, with samples at 8 and 12 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: n/a the 2 zinc capsule dosages (25 and 40 mg) will be compounded to look identical
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose 1: Zinc 25 mg/day (Experimental): 25 mg of zinc as zinc gluconate taken orally once a day
  Interventions: Drug: 25 mg/day zinc
- Dose 2: Zinc 40 mg/day (Experimental): 40 mg of zinc as zinc gluconate taken orally once a day
  Interventions: Drug: 40 mg/day zinc

INTERVENTIONS:
Drug: 25 mg/day zinc — 25 mg of zinc as zinc gluconate taken orally once a day
  Arms: Dose 1: Zinc 25 mg/day
Drug: 40 mg/day zinc — 40 mg of zinc as zinc gluconate taken orally once a day
  Arms: Dose 2: Zinc 40 mg/day

SUMMARY:
The goal of this short term prospective Phase II study is to compare the effects of two alternate daily doses of zinc (25 and 40 mg/day) in 34 randomly assigned homozygous Sickle Cell Disease (SCD-SS) patients aged 15-40 years old. The main question it aims to answer is: Which biomarkers are most responsive to zinc supplementation, and what is the maximum tolerated zinc dose that induces the desired changes in biomarkers of bone turnover? Participants will be recruited from 6 American Society Hematology Research Collaborative SCD Centers. Eligible SCD subjects will be invited to participate in the 16-week study, involving 2 baseline blood draws 4 weeks apart, followed by a 12-week zinc intervention. The findings from this study will be used to determine the dosage of zinc to be used in a larger, future study on the long term impact of zinc supplementation on bone health in SCD-SS.

DETAILED DESCRIPTION:
The investigators propose a two-arm, double-blinded, Phase II study comparing the effects of two different daily doses of zinc (25 and 40 mg/day) in 34 patients with SCD-SS aged 15-40 years old, randomly assigned to either group. The aim of the study is to determine the maximum tolerated zinc dose that induces desired changes in rates of bone formation and resorption. The findings from this study will function as preliminary data for a future randomized clinical trial and provide a novel characterization of bone marker response to short term zinc supplementation in SCD that has not previously been described in the literature.

SCD is the most prevalent heritable disorder affecting red blood cells worldwide. It is an autosomal recessive genetic condition inherited at birth when a child receives two genes, one from each parent, coding for abnormal hemoglobin. The defective hemoglobin proteins characteristic of SCD give rise to sickle-shaped red blood cells causing serious health complications, including early onset bone morbidity. Over half of young adults with SCD have osteoporosis and are at increased risk for fracture.

Zinc, an essential trace mineral, is crucial for red cell stability, growth and bone metabolism. Zinc deficiency is reported frequently in patients with SCD and has been related to poor growth, increased vaso-occlusive crises and decreased bone density. The etiology of zinc deficiency in SCD is multifactorial, including inadequate dietary intake, increased requirements due to escalations in red cell turnover and elevated urinary losses from renal insufficiency. The investigators hypothesize that bone deficits in individuals with SCD are in part due to zinc deficiency caused by oxidative stress induced hemolysis and elevated bone turnover, and these bone defects can be ameliorated by zinc supplementation.

Studies indicate that zinc improves bone density in thalassemia, a related hemoglobinopathy (Fung, 2013). But thus far, there have not been any randomized prospective studies analyzing the impact of zinc on bone health in individuals with SCD. Although emerging studies have reported that zinc supplementation might improve growth and has the potential for reducing the number and severity of sickle-related painful events, these studies are single center, small and short term. Moreover, there are currently no therapies in SCD focused on bone morbidity, and there is much enthusiasm among individuals with SCD towards participation in a nutritional intervention. A large, multicenter, long term trial of zinc supplementation focused on disease outcomes in SCD is warranted.

In order to determine the optimal tolerated dose of zinc for implementation in a future randomized clinical trial, the investigators have proposed a short term interventional study comparing the effects of two different doses of zinc, 25 vs. 40 mg/day. Subjects will be included if they are between 15 and 40 years of age, have been diagnosed with SCD-SS and are in their steady state of health. The study is a 16-week program, involving 2 baseline blood draws 4 weeks apart, followed by a randomized 12-week zinc intervention. Over the course of the study, the change in measures of bone formation and resorption, will be compared between the usual care period (0 to 4 weeks) and the intervention period (4 to 16 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 15.0 to ≤ 40.0 years
* Diagnosis: SCD-SS or SCD-S Beta zero Thalassemia, in steady state (defined as a minimum of 2 weeks days following pain crisis)
* Male or Female

Exclusion Criteria:

* Taking any supplement containing zinc and unable/willing to stop for 3 months prior to study start
* 25-Hydroxy Vitamin D < 20 ng/mL
* On chronic transfusion therapy (defined as >8 Transfusions/year) and iron overloaded (defined as liver iron concentration > 7 mg/g OR average serum ferritin >4000 ug/L)
* Unable swallow pills or take daily supplement as instructed
* Currently participating in another investigational drug trial
* Prior diagnosis of chronic kidney disease (eGFR < 30 mL/min/1.73m2)

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Biomarker of Bone Formation (PINP) | Total 16 weeks divided into: Usual Care (0 to 4 weeks) vs. Intervention Period (4 to 16 weeks)
  Bone formation will be assessed by the change in type I procollagen n-terminal propeptide (PINP) between the usual care period (0-4 weeks) and the intervention period (4-16 weeks). These assays are competitive enzyme immunoassays using microtiter plate formats. Serum will be aliquoted and frozen at -70 until analyzed in batches.
Biomarker of Bone Resorption (CTx) | Total 16 weeks divided into: Usual Care (0 to 4 weeks) vs. Intervention Period (4 to 16 weeks)
  Bone resorption will be assessed by the change in serum cross-linked C-telopeptide of type I collagen (CTx) during usual care (0 to 4 weeks) and the intervention period (4-16 weeks). These assays are competitive enzyme immunoassays using microtiter plate formats. Serum will be aliquoted and frozen at -70 until analyzed in batches.

SECONDARY OUTCOMES:
Biomarker of Bone Formation (BSAP) | Total 16 weeks divided into: Usual Care (0 to 4 weeks) vs. Intervention Period (4 to 16 weeks)
  Bone formation will be assessed by the change in bone specific alkaline phosphatase (BSAP) between the usual care period (0-4 weeks) and the intervention period (4-16 weeks). These assays are competitive enzyme immunoassays using microtiter plate formats. Serum will be aliquoted and frozen at -70 until analyzed in batches.
Biomarker of Bone Resorption (TRAP 5b) | Total 16 weeks divided into: Usual Care (0 to 4 weeks) vs. Intervention Period (4 to 16 weeks)
  Bone resorption will be assessed by the change in tartrate resistant acid phosphatase (TRAP 5b) during usual care (0 to 4 weeks) and the intervention period (4-16 weeks). These assays are competitive enzyme immunoassays using microtiter plate formats. Serum will be aliquoted and frozen at -70 until analyzed in batches.

OTHER OUTCOMES:
Tolerability of Zinc Supplement | Total 16 weeks divided into: Usual Care (0 to 4 weeks) vs. Intervention Period (4 to 16 weeks)
  We will monitor tolerability of each dose of zinc by subject documentation of abdominal pain, cramping, nausea, vomiting, anorexia, diarrhea and headaches in daily response within the Think Zinc reminder app while supplemented with zinc (25 or 40 mg/day) compared to baseline period.
Adherence to Zinc Supplementation | Total 12 weeks during Intervention Period (4 to 16 weeks)
  We will monitor adherence to the zinc supplement (25 or 40 mg/day) through subject responses to the daily Think Zinc reminder App, as well as pill counts at the end of the 3 month supplementation period.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Fung, PhD, Principal Investigator — University of California, San Francisco
Locations (6):
- United States (6):
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Data sharing available upon request after the completion of the trial
Supporting Information: Study Protocol, SAP, ICF
Time Frame: upon completion of the trial the information will be available for 1 year

REFERENCES:
- [Background] Fung EB, Kwiatkowski JL, Huang JN, Gildengorin G, King JC, Vichinsky EP. Zinc supplementation improves bone density in patients with thalassemia: a double-blind, randomized, placebo-controlled trial. Am J Clin Nutr. 2013 Oct;98(4):960-71. doi: 10.3945/ajcn.112.049221. Epub 2013 Aug 14. PMID 23945720